CLINICAL TRIAL: NCT02476591
Title: Charge Transparency in Critical Care Practice and Its Effects on Overall Cost of Care: Physician Awareness of ICU Charge Environment: The PRICE Study
Brief Title: Charge Transparency in Critical Care Practice and Its Effects on Overall Cost of Care
Acronym: PRICE
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Adam Kingeter, Fellow, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 150722
Record Dates: First submitted 2015-06-11; First posted 2015-06-19 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Intensive Care
Keywords: Resource utilization; intensive care unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Charge transparency: Providers with access to charge transparency as displayed via a dashboard with patient specific charge data for a given ICU stay
  Interventions: Behavioral: Charge Transparency
- Without charge transparency: Providers without access to patient specific charge data

INTERVENTIONS:
Behavioral: Charge Transparency — Providers caring for patients in the "Charge Transparency" cohort will be given access to patient specific charge data on a daily basis via an interactive dashboard which allows for full charge transparency to patients admitted to the Vanderbilt ICUs
  Groups: Charge transparency

SUMMARY:
To investigate the effects of the availability of daily patient-related charges on ordering patterns of health care ordering providers and cost containment in the Intensive Care Unit (ICU) setting.

DETAILED DESCRIPTION:
Ordering providers include resident, fellow and attending physicians, as well as mid level providers such as Nurse Practitioners (NP's) and Physician Assistants (PA's). The investigators have developed a dashboard that displays both daily and cumulative charges related to laboratory, pharmacy, radiology, and other services for all patients admitted to Vanderbilt ICU's. Using this dashboard an ICU ordering provider is able to see not only the total daily charges for the previous 24 hours, but also the sum of all charges for that patient's current ICU admission. In addition, a "snapshot" overview tab is available for each patient that displays a day by day trend of the overall charges of the ICU stay for the patient, top 5 most expensive lab/radiology/pharmacy charges, previous 24 hour charges, and the total ICU number of chest x-ray, Complete Blood Count (CBC), Basic Metabolic Panel (BMP), Electrocardiogram (EKG), and Arterial Blood Gas (ABG) charges to the patient. The ordering provider is able to query the database of the dashboard for information regarding individual laboratory and drug charges, as well as view trajectory of total charges for a given patient. This dashboard allows for unprecedented transparency regarding the cost of care for patients in an ICU. Patients are identified in the dashboard by Medical Record Number (MRN), ICU bed, and initials only so as to protect their identity.

AIM 1: To evaluate the effects of introducing charge transparency to ordering providers via a charge dashboard and associated printed synopsis on average charge per patient per day in the Vanderbilt ICUs.

We intend to study the effect of charge transparency to ordering providers on average charge per patient per day by conducting a prospective, self-controlled by unit, multiple cross-over trial. We will divide the study period into four 12-week blocks with two blocks of "charge transparency" and two blocks of "no transparency." Each unit will be assigned to alternating blocks of "transparency" and "no transparency" during the study with each unit on the same schedule so as to prevent cross contamination.

For months during which access is granted, all ordering providers in the study ICU will be granted access to the ICU charge dashboard following a brief orientation. In addition a password protected, unit specific iPad will be provided to each study unit. The iPad will enable point of care access to the patient specific snapshot information, as well as easily incorporate the dashboard information into clinical care.

AIM 2: To evaluate the effects of utilization of a charge dashboard on ordering patterns of providers and cost containment in the Vanderbilt ICUs.

In addition to studying the effect of charge transparency on patient ICU charges, we also intend to study the effect of charge transparency on resource utilization, namely routine laboratory and radiology tests. As surrogate markers for routine laboratory utilization we will measure average number of Comprehensive Blood Count (CBC) and Basic Metabolic Panel (BMP) tests per patient per day, and as surrogate markers for routine radiology utilization we will use average number of chest x-rays per patient per day.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the Vanderbilt University Medical Center Cardiovascular, Surgical, Burn, Medical and Neuroscience ICUs will be included

Exclusion Criteria:

* There are no exclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the Vanderbilt University Medical Center Cardiovascular, Surgical, Burn, Medical and Neuroscience ICUs will be included
Sampling Method: Non-Probability Sample
Enrollment: 10720 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2016-10-03 (Actual); Study Completion 2016-10-03 (Actual)

PRIMARY OUTCOMES:
Average charge per patient per day ($) | 12 week block
  Sum hospital charges for each study unit during the 12 week block will be divided by total number of patients admitted to the study unit during that time, and again by 84 days to obtain average charge per patient per day in the ICU during the study period for each cohort.

SECONDARY OUTCOMES:
Average number of Basic Metabolic Panels per patient per day | 12 week blocks
  Sum total of basic metabolic panels for each study unit during the 12 week block will be divided by total number of patients admitted to the study unit during that time, and again by 84 days to obtain average number of basic metabolic panels per patient per day in the ICU during the study period for each cohort.
Average number of complete blood counts per patient per day | 12 weeks
  Sum total of complete blood counts for each study unit during the 12 week block will be divided by total number of patients admitted to the study unit during that time, and again by 84 days to obtain average number of complete blood counts per patient per day in the ICU during the study period for each cohort.
Average number of chest x-rays per patient per day | 12 weeks
  Sum total of portable chest x-rays for each study unit during the 12 week block will be divided by total number of patients admitted to the study unit during that time, and again by 84 days to obtain average number of chest x-rays per patient per day in the ICU during the study period for each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Kingeter, MD, Principal Investigator — Vanderbilt University Medical Center